CLINICAL TRIAL: NCT00743301
Title: Effects of Palm Olein Versus Olive Oil on Blood Lipids, Lipoproteins and Novel Risk Markers of Cardiovascular Disease
Brief Title: The Effect of Palm Olein, Olive Oil and Lard and on Risk Markers of Cardiovascular Disease
Acronym: A305
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Tine Tholstrup, Dpt Human Nutrition, University of Copenhagen, Denmark
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: HB2008-056
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Last update posted 2008-08-28 (Estimated); Status verified 2008-08

CONDITIONS: Cardiovascular Disease; Metabolic Syndrome
Keywords: CVD; Palm olein; Olive oil; Lard; healthy men; metabolic syndrome; Risk of cardiovascular disease and metabolic syndrome
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Syndrome | interventions — lard

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Olive oil (Active Comparator)
  Interventions: Other: Palm olein vs olive oil and lard
- Palm olein (Experimental)
  Interventions: Other: Palm olein vs olive oil and lard
- Lard (Active Comparator)
  Interventions: Other: Palm olein vs olive oil and lard

INTERVENTIONS:
Other: Palm olein vs olive oil and lard — 17E% from test fat is incorporated into three rolls and a piece of cake

SUMMARY:
The aim of this study is to compare the effects of a diet rich in palm olein, a fraction of palm oil, to a diet rich in olive oil and a diet rich in Danish lard on plasma total-, LDL and HDL cholesterol as well as triacylglycerol (TAG), fasting insulin and glucose, C reactive protein and plasminogen activator inhibitor 1 in healthy men. The investigators hypothesis is that palm olein and olive oil will have the same effect on plasma total cholesterol, LDL- and HDL concentration and maybe also on the secondary outcome parameters that are related to cardiovascular disease risk. This may be caused by the differences in the sn-positioning of palmitic acid in palm olein. This difference may cause the palmitic acid in palm olein to be more prone to soap formations and excretion than palmitic acid from other sources, e.g. lard.

This study is a double blinded, randomized, controlled 3 x 3 week crossover intervention study, without washout periods. The participants receive the three test foods in random order, decided by draw of lots. Blood samples are drawn in duplicate (on two following days) before and after each dietary period.

ELIGIBILITY:
Inclusion Criteria:

1. All participants must give their informed consent in writing, after having received oral and written information about the study
2. Age: 18-65 y
3. BMI: 18.5 - 30 mg/m2
4. Men
5. Healthy (no known diseases, incl. hypertension, hypercholesterolemia, diabetes and psoriasis)
6. No use of dietary supplements or blood donations two month prior to and during the intervention

Exclusion Criteria:

1. Current or previously cardiovascular disease
2. Diabetes Mellitus or other severe chronic disease, including severe allergies and psoriasis
3. Hypertension
4. Known or suspected abuse of alcohol, drugs or medication
5. Own request: all participants have the right to withdraw from the intervention at any given time without explanation
6. Compliance: participants may be excluded from the intervention if they do not follow the study guidelines
7. Side effects (There are no side effects expected in this study since all test fats are commercial available and use in households world wide)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-02 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
total, HDL, LDL cholesterol and triacylglycerol | before and after each type of dietary fat

SECONDARY OUTCOMES:
fasting insulin and glucose, c reactive protein and plasminogen activator inhibitor 1 | befoer and after each dietary test fat

CONTACTS AND LOCATIONS:
Overall Officials: Tine Tholstrup, PhD, Principal Investigator — Department of Human Nutrition, University of Copenhagen
Locations (1):
- Department of Human Nutrition, Frederiksberg, Denmark

REFERENCES:
- [Derived] Tholstrup T, Hjerpsted J, Raff M. Palm olein increases plasma cholesterol moderately compared with olive oil in healthy individuals. Am J Clin Nutr. 2011 Dec;94(6):1426-32. doi: 10.3945/ajcn.111.018846. Epub 2011 Nov 9. PMID 22071711